CLINICAL TRIAL: NCT02901899
Title: An Open Label Phase II Trial of Guadecitabine and Pembrolizumab in Platinum Resistant Recurrent Ovarian Cancer
Brief Title: Guadecitabine and Pembrolizumab in Treating Patients With Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Astex Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniela Matei, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16G03; STU00203494 (CTRP (Clinical Trial Reporting Program)); NU 16G03 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01296 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — guadecitabine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (guadecitabine, pembrolizumab) (Experimental): Patients receive guadecitabine SC on days 1-4 and pembrolizumab IV over 30 minutes on day 5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Guadecitabine; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI-110
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
The purpose of this study is to look at how patients respond to treatment with guadecitabine and pembrolizumab. The researchers will also be looking at the amount of time it takes for cancer to get worse when participants take the study drugs. All participants will be treated with guadecitabine and pembrolizumab. Guadecitabine interferes with the cancer cells' DNA and can increase the production of certain proteins, making cancer cells more recognizable by the immune system. Pembrolizumab helps your immune system to kill cancer cells. Thus the combination of guadecitabine and pembrolizumab may increase the ability of the immune system to eliminate cancer cells. Researchers want to find out whether the combination of guadecitabine and pembrolizumab is effective in treating ovarian cancer that has not responded to traditional chemotherapy. Participants will keep receiving treatment until their cancer gets worse, they have side effects, or they decide they don't want to receive the treatment anymore. After stopping treatment, the study doctor will watch participants for side effects and follow their condition every 6-12 weeks. The study aims to keep track of participants' medical conditions for the rest of their lives. This helps us look at the long-term effects of the study drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure objective response rate (RR) to guadecitabine and pembrolizumab in subjects with recurrent platinum resistant ovarian cancer (OC).

SECONDARY OBJECTIVES:

I. Measure progression free survival (PFS) for the combination of guadecitabine and pembrolizumab.

II. Progression free survival (PFS). III. Measure clinical benefit rate (CBR) for the combination of guadecitabine and pembrolizumab.

IV. Measure toxicity profiles to the combination of guadecitabine and pembrolizumab.

TERTIARY OBJECTIVES:

I. NY-ESO-1 and MAGE antigens' promoter methylation (pyrosequencing) and messenger ribonucleic acid (mRNA) expression levels (quantitative reverse transcriptase-polymerase chain reaction [RT-PCR]) will be measured before and after treatment in deoxyribonucleic acid (DNA) (plasma and/or tumor biopsies) and ribonucleic acid (RNA) (tumor biopsies), respectively.

II. Cytokine response (IFN gamma IL2, IL6, IL10, TNF alpha) will be measured in plasma by enzyme-linked immunosorbent assay (ELISA).

III. Measure LINE 1 methylation in DNA extracted from peripheral blood mononuclear cells (PBMCs) (measured on days 1 and 5 of cycles 1 and 2).

IV. Expression of the PD-L1 ligand will be measured by immunohistochemistry (IHC) in archival tumors.

V. Tumor infiltrating lymphocytes (TILs) will be quantified in tumor biopsies before and after treatment (IHC).

OUTLINE:

Patients receive guadecitabine subcutaneously (SC) on days 1-4 and pembrolizumab intravenously (IV) over 30 minutes on day 5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 6 weeks for 1 year, and then every 9 weeks and, once a subject experiences confirmed disease progression or starts a new anticancer therapy, every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or cytological evidence/confirmation of recurrent epithelial ovarian cancer, primary peritoneal carcinomatosis, or fallopian tube cancer
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 within 28 days prior to registration
* Prior therapy allowed:

  * At least one and no more than 3 platinum based chemotherapy regimens
  * Up to 2 non-platinum, cytotoxic regimen
  * There is no limit on use of prior biological therapies (hormonal or targeted therapy)
  * NOTE: Prior immunotherapy is not allowed
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG), performance status of 0-1 within 14 days prior to registration
* Demonstrate adequate organ function as defined below; all screening labs to be obtained within 14 days prior to treatment initiation:
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (without transfusion or growth factor support/erythropoietin [EPO] dependency)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Be willing to allow the use of archival formalin-fixed paraffin-embedded tumor tissue for correlative analyses

  * Note: The archived tumor tissue specimens may be from prior surgery or from prior diagnostic biopsy of primary or metastatic tumor specimen; unavailability of archived tissue will not render subject ineligible for study
* Be willing and able to undergo a core or excisional tumor biopsy according to institutional standards (guided visually or by computed tomography [CT] or ultrasound), paracentesis, or thoracentesis for tumor cells

  * Note: This is to be done prior to treatment at cycle 1 day 1 (C1D1) and post-treatment (cycle 2 day 8), if this is clinically and safely feasible to do so; this will allow the use of this freshly obtained tissue for correlative analyses in the study
* Females of child-bearing potential (FOCBP) must agree to use adequate contraception prior to registration, for the duration of study participation, and for 120 days following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative pregnancy test within 7 days prior to registration on study
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * NOTE: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * NOTE: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has had a prior anti-cancer monoclonal antibody (mAb) within 28 days prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days registration
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days prior to registration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent; please contact the principal investigator for further clarification if needed
* Hypersensitivity to pembrolizumab or any of its excipients
* Has a known history of active TB (Bacillus tuberculosis)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) infection
* Has a known history of hepatitis B and/or hepatitis C infection
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy within 3 days of registration (NOTE: except for uncomplicated urinary tract infection [UTI])
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Female patients who are pregnant or nursing, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment; subjects should not breast feed within 120 days of completing the trial
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific subject

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois

REFERENCES:
- [Derived] Chen S, Xie P, Cowan M, Huang H, Cardenas H, Keathley R, Tanner EJ, Fleming GF, Moroney JW, Pant A, Akasha AM, Davuluri RV, Kocherginsky M, Zhang B, Matei D. Epigenetic priming enhances antitumor immunity in platinum-resistant ovarian cancer. J Clin Invest. 2022 Jul 15;132(14):e158800. doi: 10.1172/JCI158800. PMID 35671108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual May 23, 2016 with the first patient being treated on study November 14, 2016. The study was suspended January 30 2017 pending completion of safety run in and data review, reopening March 22 2017. The study closed to further accrual November 25 2019 with accrual being considered to be met.
Groups:
- Treatment (Guadecitabine, Pembrolizumab): Patients receive guadecitabine as a subcutaneous injection on Days 1-4 and pembrolizumab as a IV infusion over 30 minutes on Day 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Reached 1st Response Assessment
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Started | 45
Registered | 45
Started Treatment | 43
Attempted 2 Cycles of Treatment/Reached First Response | 37
Completed | 37
Not Completed | 8
Period: Continued Treatment After 1st Response
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Started (Treatment may continue in the absence of disease progression, unacceptable toxicity, death and withdrawal from the study.) | 37
Went on to Start Cycle 3 | 21
Completed | 21
Not Completed | 16
Period: Follow up
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Started (Follow up continues until death, withdrawal of consent or the end of the study, whichever comes first.) | 43 (All patients who receive at least one dose of study drug go into the follow up period.)
Completed | 27
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 61 [34 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 36
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Using RECIST 1.1
Description: Objective response rate (ORR) is defined as the number of patients who's best response is complete response plus those with partial response. Imaging scans will be assessed using RECIST 1.1 to measure ORR to guadecitabine and pembrolizumab in patients with recurrent platinum resistant Ovarian Cancer.
  In general the following definitions apply Complete Response - Disappearance of all lesions Partial Response - At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessed from start of treatment and during treatment for up to 38 cycles where 1 cycle equals 21 days (maximum number of cycles that any patient attempted)
Population: Per protocol patients need to complete at least 2 cycles of treatment to be evaluable for this endpoint.
Measure: Number; unit: patients
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Number analyzed (Participants) | 38
patients | 3

2. Secondary Outcome: Objective Response Rate (ORR) Using Immune Related Response Criteria (irRC)
Description: Objective response rate (ORR) is defined as the number of complete responders and partial responders divided by the patient population evaluable for response. Imaging scans will be assessed using the using the Immune Related Response Criteria (irRC) to measure ORR to guadecitabine and pembrolizumab in patients with recurrent platinum resistant Ovarian Cancer.
Time Frame: Up to 3 years
Population: This endpoint was not analyzed because the data required for analysis was not collected.
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as the duration of time from treatment start to time of progression or death, whichever occurs first. The median PFS value (in months) is reported here. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 3 years
Population: Only patients that completed at least 1 cycle of treatment were analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Number analyzed (Participants) | 43
months | 1.74 [1.25 to 2.76]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the number of patients who's best response is complete response, plus those with partial response plus those with stable disease as evaluated using imagining scans and assessed by RECIST 1.1 and received at least 6 cycles of treatment.
  Complete Response - Disappearance of all lesions Partial Response - At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease - Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study
Time Frame: as for outcome 1
Population: Patient must receive at least 2 cycles of treatment to be evaluable for this endpoint
Measure: Number; unit: patients
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Number analyzed (Participants) | 35
patients | 9

5. Secondary Outcome: Incidence of Adverse Events
Description: Assess the toxicity of guadecitabine and pembrolizumab by measuring the number, type, grade, severity, and frequency of adverse events according to the National Cancer Institute Common Terminology Criteria Adverse events (AE) (CTCAE) v 4.03. Those that were determined to be at least possibly related to study drugs are reported per drug (guadecitabine and pembrolizumab). Number of related Serious Adverse Events (SAEs) is also reported
Time Frame: Assessed from start of treatment and during treatment for up to 38 cycles and up to 90 days post last dose where 1 cycle equals 21 days (maximum number of cycles that any patient attempted)
Measure: Number; unit: participants
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
Number analyzed (Participants) | 43
participants
  Related to Guadecitabine : All AEs | 41
  Related to Guadecitabine : AEs graded 1-2 | 40
  Related to Guadecitabine : AEs graded 3-4 | 23
  Related to Guadecitabine : SAEs | 3
  Related to Pembrolizumab : All AEs | 33
  Related to Pembrolizumab : AEs graded 1-2 | 32
  Related to Pembrolizumab : AEs graded 3-4 | 9
  Related to Pembrolizumab : SAEs | 6

ADVERSE EVENTS:
Time Frame: Patients are assessed for adverse events (AE) from the start of the treatment, every cycle and for 30 days post last dose of treatment (up to 90 days post last dose of treatment) for up to a maximum of 38 cycles where cycles are 21 days in length, up to a total of 3 years
Description: Patients registered to the study who did not start treatment were not assessed for AEs and not included. There were a total of 29 SAEs but some contained multiple event terms. Each SAE event term is included here.
Arm/Group | Treatment (Guadecitabine, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 29/43
Serious Adverse Events (participants affected / at risk) | 18/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Guadecitabine, Pembrolizumab) (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Guadecitabine, Pembrolizumab) (N=43)
Anemia (Blood and lymphatic system disorders) | 22 (55)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 13 (20)
Ascites (Gastrointestinal disorders) | 4 (5)
Bloating (Gastrointestinal disorders) | 6 (8)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 12 (17)
Diarrhea (Gastrointestinal disorders) | 12 (18)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (28)
Obstruction gastric (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 11 (15)
Chills (General disorders) | 7 (7)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 19 (22)
Fever (General disorders) | 7 (7)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Injection site reaction (General disorders) | 12 (23)
Irritability (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Tooth infection (Infections and infestations) | 3 (4)
Upper respiratory infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 5 (6)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 4 (6)
Alanine aminotransferase increased (Investigations) | 4 (7)
Alkaline phosphatase increased (Investigations) | 10 (23)
Aspartate aminotransferase increased (Investigations) | 8 (12)
Blood bilirubin increased (Investigations) | 3 (4)
Creatinine increased (Investigations) | 3 (5)
INR increased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 9 (13)
Lymphocyte count decreased (Investigations) | 28 (83)
Neutrophil count decreased (Investigations) | 23 (49)
Platelet count decreased (Investigations) | 6 (13)
Weight loss (Investigations) | 7 (12)
White blood cell decreased (Investigations) | 29 (76)
Anorexia (Metabolism and nutrition disorders) | 14 (17)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 8 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 8 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Concentration impairment (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 6 (6)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Confusion (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 4 (4)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 4 (5)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (3)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (10)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (8)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 3 (3)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 14 (73)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT02901899/Prot_SAP_000.pdf